CLINICAL TRIAL: NCT04033614
Title: Fasciotens to Treat an Open Abdomen - a Prospective Cohort Study
Acronym: Fasciotens
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Collaborators: Fasciotens GmbH (Unknown)
Responsible Party: Principal Investigator, Dr. Roman Marius Eickhoff, Specialist in surgery, RWTH Aachen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-019
Record Dates: First submitted 2019-07-18; First posted 2019-07-26 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Abdominal Compartment Syndrome; Pancreatitis,Acute Necrotizing; Intraabdominal Hypertension; Peritonitis
Keywords: Laparotomy, open abdomen, fascia, retraction, intraabdominal oedema
MeSH Terms: conditions — Intra-Abdominal Hypertension; Pancreatitis, Acute Necrotizing; Peritonitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Laparostoma (Experimental): Patients needing a laparostoma will be treated with the fasciotens abdomen device. The distance between the fasciae will be measured frequently using a ruler.
  12 months after the treatment an ultrasound measurement will be performed to assess hernia formation
  Interventions: Device: Fasciotens-Abdomen

INTERVENTIONS:
Device: Fasciotens-Abdomen — The basic principle of Fasciotens Abdomen is the ventrally directed pulling force on the two fascial edges via an external device with support on the thorax and pelvis. A commercially available resorbable surgical mesh is sewn into the fascia margin. Commercial surgical sutures attached to this net are then attached to a height-adjustable suspension, which is connected to an external support on the thorax and pelvis. This ensures continuous traction to the two fascial edges. The remaining wound surface can then be treated with conventional dressing material.

SUMMARY:
The open abdomen can occur as a result of various diseases. After infections of the abdomen, compartment syndromes or traumata, it is essential for survival (1). This condition of the open abdomen lasts from days to months. Within a very short time, the fascia and abdominal wall structures retract in such a way that direct abdominal closure is often impossible. In addition, there is a pronounced intraabdominal oedema, which additionally increases the space required by the abdominal organs. Therefore, it is clinically indispensable to increase the space of the intraabdominal organs in this life-threatening situation. After the laparotomy (opening of the abdomen) has been performed, it is therefore not closed. However, the natural traction on the abdominal wall, in particular on the fascia, the attached musculature as well as skin and subcutis, no longer exists in this situation. As a result, these structures retract over the period of the existing laparostoma.

In the present study, the CE-certified medical device Fasciotens Abdomen will be used to prove the functionality of this device and the user feasibility.

The basic principle of Fasciotens Abdomen is the ventrally directed pulling force on the two fascial edges via an external device with support on the thorax and pelvis. The possibility to apply a traction to the fascia from the moment of opening the abdomen without reducing the intraabdominal space is absolutely new and the rationale of this technique. The objective of this study is to prove the obvious prevention of fascial retraction through the Fasciotens Abdomen device.

DETAILED DESCRIPTION:
The open abdomen can occur as a result of various diseases. After infections of the abdomen, compartment syndromes or traumata, it is essential for survival (1). This condition of the open abdomen lasts from days to months. Within a very short time, the fasciae and abdominal wall structures retract in such a way that direct abdominal closure is often impossible. In addition, there is a pronounced intraabdominal oedema, which additionally increases the space required by the abdominal organs. Therefore, it is clinically indispensable to increase the space of the intraabdominal organs in this life-threatening situation. After the laparotomy (opening of the abdomen) has been performed, it is therefore not closed. However, the natural traction on the abdominal wall, in particular on the fascia, the attached musculature as well as skin and subcutis, no longer exists in this situation. As a result, these structures retract over the period of the existing laparostoma.

The current state of the art is the treatment of the open abdomen using low-pressure therapy or other temporary abdominal wall closure. The most common method is pure vacuum dressing on the abdominal wall wound and the abdominal organs (2, 3). However, traction to the edges of the fascia is only possible after the intraabominal increase in volume and pressure has decreased. All previously described methods for temporary abdominal wall closure cannot counteract abdominal wall retraction and can only begin with a pull on the already retracted fascia after normalization of the abdominal volume.

The later abdominal closure then often requires alloplastic materials or results in a defect healing as abdominal wall hernia (4, 5). The temporal extension of the open abdomen is also associated with intestinal adhesions, formation of intestinal fistula and loss of abdominal volume (6-12). Mortality of the open abdomen is 12-40%, with septic genesis associated with higher mortality (1). In addition, reocclusion should be sought at an early stage. Trauma patients with a re-closure within 48 hours show a more favourable course of disease, a lower complication rate and lower mortality (13-15). The retraction of the abdominal wall and the later often impossible abdominal closure are the main problems in the treatment of these seriously ill patients. This problem, which has not yet been solved, is the reason for the development of this new technique.

In the present study, the CE-certified medical device Fasciotens Abdomen will be used to prove the functionality of this device and the user feasibilty.

The basic principle of Fasciotens Abdomen is the ventrally directed pulling force on the two fascial edges via an external device with support on the thorax and pelvis. A commercially available resorbable surgical mesh is sewn into the fascia margin, which would also have been used without the Fasciotens system. Commercial surgical sutures attached to this net are then attached to a height-adjustable suspension, which is connected to an external support on the thorax and pelvis. This ensures continuous traction to the two fascial edges. This counteracts the natural muscle pull of the abdominal muscles and thus the retraction of the abdominal wall to both sides laterally. At the same time the abdomen is still open preventing necrosis of the abdominal organs. The remaining wound surface can then be treated with conventional dressing material.

The possibility to apply a traction to the fascia from the moment of opening the abdomen without reducing the intraabdominal space is absolutely new and the rationale of this technique. The objective of this study is to prove the obvious prevention of fascial retraction through the Fasciotens Abdomen device.

ELIGIBILITY:
Inclusion Criteria:

* Laparostoma with a resorbable net and planned or necessary "second look" operation.
* Age of majority
* Signed informed consent form or in the case of patients unable to give consent, signature from the authorised representative/legal carevier or consultant.

Exclusion Criteria for the period of use of the Fasciotens Abdomen device:

* Pregnancy or breast-feeding at the time of inclusion into the study
* A Moribund patient with a life expectancy of less than 24 hours despite laparostomy
* Unstable thorax or known severe skeletal instability which impaires the use of the fasciotens abdomen device.
* Open wounds or infections at the potential contact points of the Fasciotens abdomen device
* Known cardiac insufficiency with ejection fraction less than 35%
* Patients with lung failure (ARDS) and the need for abdominal positioning within the next 24h

Exclusion criteria for the entire duration of the study:

* Persons who are accommodated in a mental hospital or an insititution on official or judicial instruction
* Persons who are dependent on or have an employment relationship with the principal investigator
* Other conditions which, at the judgement of the investigator, militate against the use of the investigational product
* Minority

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-08-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Closure rate of the abdominal wall fascia | Up to 24 weeks
  The primary endpoint of the study is the closure rate of the fascia.

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik für Allgemein-, Viszeral- und Transplantationschirurgie, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bruhin A, Ferreira F, Chariker M, Smith J, Runkel N. Systematic review and evidence based recommendations for the use of negative pressure wound therapy in the open abdomen. Int J Surg. 2014 Oct;12(10):1105-14. doi: 10.1016/j.ijsu.2014.08.396. Epub 2014 Aug 28. PMID 25174789
- [Background] Quyn AJ, Johnston C, Hall D, Chambers A, Arapova N, Ogston S, Amin AI. The open abdomen and temporary abdominal closure systems--historical evolution and systematic review. Colorectal Dis. 2012 Aug;14(8):e429-38. doi: 10.1111/j.1463-1318.2012.03045.x. PMID 22487141
- [Background] Roberts DJ, Zygun DA, Grendar J, Ball CG, Robertson HL, Ouellet JF, Cheatham ML, Kirkpatrick AW. Negative-pressure wound therapy for critically ill adults with open abdominal wounds: a systematic review. J Trauma Acute Care Surg. 2012 Sep;73(3):629-39. doi: 10.1097/TA.0b013e31825c130e. PMID 22929494
- [Background] Carlson GL, Patrick H, Amin AI, McPherson G, MacLennan G, Afolabi E, Mowatt G, Campbell B. Management of the open abdomen: a national study of clinical outcome and safety of negative pressure wound therapy. Ann Surg. 2013 Jun;257(6):1154-9. doi: 10.1097/SLA.0b013e31828b8bc8. PMID 23478532
- [Background] Cheatham ML, Demetriades D, Fabian TC, Kaplan MJ, Miles WS, Schreiber MA, Holcomb JB, Bochicchio G, Sarani B, Rotondo MF. Prospective study examining clinical outcomes associated with a negative pressure wound therapy system and Barker's vacuum packing technique. World J Surg. 2013 Sep;37(9):2018-30. doi: 10.1007/s00268-013-2080-z. PMID 23674252
- [Background] Cheatham ML, Safcsak K. Is the evolving management of intra-abdominal hypertension and abdominal compartment syndrome improving survival? Crit Care Med. 2010 Feb;38(2):402-7. doi: 10.1097/ccm.0b013e3181b9e9b1. PMID 20095067
- [Background] Miller RS, Morris JA Jr, Diaz JJ Jr, Herring MB, May AK. Complications after 344 damage-control open celiotomies. J Trauma. 2005 Dec;59(6):1365-71; discussion 1371-4. doi: 10.1097/01.ta.0000196004.49422.af. PMID 16394910
- [Background] Vidal MG, Ruiz Weisser J, Gonzalez F, Toro MA, Loudet C, Balasini C, Canales H, Reina R, Estenssoro E. Incidence and clinical effects of intra-abdominal hypertension in critically ill patients. Crit Care Med. 2008 Jun;36(6):1823-31. doi: 10.1097/CCM.0b013e31817c7a4d. PMID 18520642
- [Background] Raeburn CD, Moore EE, Biffl WL, Johnson JL, Meldrum DR, Offner PJ, Franciose RJ, Burch JM. The abdominal compartment syndrome is a morbid complication of postinjury damage control surgery. Am J Surg. 2001 Dec;182(6):542-6. doi: 10.1016/s0002-9610(01)00821-2. PMID 11839314
- [Background] Barker DE, Kaufman HJ, Smith LA, Ciraulo DL, Richart CL, Burns RP. Vacuum pack technique of temporary abdominal closure: a 7-year experience with 112 patients. J Trauma. 2000 Feb;48(2):201-6; discussion 206-7. doi: 10.1097/00005373-200002000-00001. PMID 10697075
- [Background] Bee TK, Croce MA, Magnotti LJ, Zarzaur BL, Maish GO 3rd, Minard G, Schroeppel TJ, Fabian TC. Temporary abdominal closure techniques: a prospective randomized trial comparing polyglactin 910 mesh and vacuum-assisted closure. J Trauma. 2008 Aug;65(2):337-42; discussion 342-4. doi: 10.1097/TA.0b013e31817fa451. PMID 18695468
- [Background] De Waele JJ, Leppaniemi AK. Temporary abdominal closure techniques. Am Surg. 2011 Jul;77 Suppl 1:S46-50. PMID 21944452
- [Background] Hatch QM, Osterhout LM, Podbielski J, Kozar RA, Wade CE, Holcomb JB, Cotton BA. Impact of closure at the first take back: complication burden and potential overutilization of damage control laparotomy. J Trauma. 2011 Dec;71(6):1503-11. doi: 10.1097/TA.0b013e31823cd78d. PMID 22182860
- [Background] Burlew CC, Moore EE, Biffl WL, Bensard DD, Johnson JL, Barnett CC. One hundred percent fascial approximation can be achieved in the postinjury open abdomen with a sequential closure protocol. J Trauma Acute Care Surg. 2012 Jan;72(1):235-41. doi: 10.1097/TA.0b013e318236b319. PMID 22310132
- [Background] Dubose JJ, Scalea TM, Holcomb JB, Shrestha B, Okoye O, Inaba K, Bee TK, Fabian TC, Whelan J, Ivatury RR; AAST Open Abdomen Study Group. Open abdominal management after damage-control laparotomy for trauma: a prospective observational American Association for the Surgery of Trauma multicenter study. J Trauma Acute Care Surg. 2013 Jan;74(1):113-20; discussion 1120-2. doi: 10.1097/TA.0b013e31827891ce. PMID 23271085
- [Background] Lambertz A, Mihatsch C, Roth A, Kalverkamp S, Eickhoff R, Neumann UP, Klink CD, Junge K. Fascial closure after open abdomen: initial indication and early revisions are decisive factors--a retrospective cohort study. Int J Surg. 2015 Jan;13:12-16. doi: 10.1016/j.ijsu.2014.11.025. Epub 2014 Nov 25. PMID 25447607